CLINICAL TRIAL: NCT00188084
Title: Analysis of Four Biological Parameters at Diagnosis of Adult Acute Lymphoblastic Leukaemia: DNA Index, Percentage of Cells in S-Phase, CD45 Fluorescence Index, and Protein P16: Prognostic Study in Patients Enrolled in a Multicentric Trial
Brief Title: Description and Prognostic Evaluation of Four Biological Parameters of Blast Cells in Adult Acute Lymphoblastic Leukemia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Angers (Other Government)
Collaborators: French Innovative Leukemia Organisation (Other)
Other Study IDs: PHRC03-02; GOELAMS 271-003
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2005-10-28 (Estimated); Status verified 2005-09

CONDITIONS: Adult Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Ploidies; S Phase

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

INTERVENTIONS:
Procedure: DNA Index
Procedure: S-Phase%
Procedure: CD45 expression
Procedure: P16 metabolic way

SUMMARY:
Adult acute lymphoblastic leukemia treatment approaches relie on risk stratification, including cytogenetics. We want to study at diagnosis several blast cells parameters on frozen samples of GRAALL protocols enrolled patients:

1. A CD45-DNA double staining analysed by flow cytometry will allow mesurement for each blastic clone of DNA ploidy, percentage of cells in S-phase, CD45 fluorescence index.
2. The proteine P16 metabolic way, involved in cell cycle regulation, will be studied by Western Blot analysis.

The comparison between these parameters, and main haematological data, will be followed by a prognostic analysis, based on blast corticosensibility in vivo, chimiosensibility, complete remission, and survival.

Combination of the studied parameters will allow to appreciate a clonal diversity. This will help to predict, at diagnosis, high probability of resistance to treatment.

ELIGIBILITY:
Inclusion Criteria:

* All GRAALL 2003 and 2005 enrolled patients with available frozen blast cells

Exclusion Criteria:

* None

Ages: 15 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 400
Dates: Start 2003-11; Study Completion 2005-09

CONTACTS AND LOCATIONS:
Overall Officials: Laurence M Baranger, MD, Principal Investigator — University Hospital, Angers
Locations (1):
- CRLCC Centre Paul Papin, Angers, France